CLINICAL TRIAL: NCT03485261
Title: Sexual Dysfunctions in Female Patients With Chronic Kidney Disease
Brief Title: Female Sexual Dysfunctions in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Mohamed, eamohamed, Assiut University
Other Study IDs: FSDCKD
Record Dates: First submitted 2018-03-27; First posted 2018-04-02 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: patient group include 50 female patients with chronic renal failure (eGFR <15ml/min/1.7m2 )
- Group B: the control group including 50 healthy females age matched with the patient group

SUMMARY:
A myriad of sexual problems affect men and women with chronic kidney disease (CKD), including decreased libido, erectile dysfunction, dysmenorrhea, and infertility. Menstrual abnormalities are common in CKD and many women are an-ovulatory.

Sexual dysfunction in CKD is multifactorial including hormonal alterations along with vascular, neurologic, psychogenic, and other factors, such as medications, contribute to the development of sexual dysfunction. Sexual dysfunction in females is mainly due to hormonal factors and manifests mainly as menstrual irregularities, amenorrhea, lack of vaginal lubrication, and failure to conceive.

DETAILED DESCRIPTION:
The study will be conducted on 100 female patients divided in to two equal group:

1. Group A: The patient group include 50 female patients with chronic renal failure (eGFR <15ml/min/1.7m2 )
2. Group B: The control group including 50 healthy females age matched with the patient group.

The Female Sexual Function Index (FSFI) will be used to assess sexual function. This index includes 19 questions related to 6 parameters: sexual desire, sexual arousal, lubrication, orgasm, sexual satisfaction and dyspareunia. A face-to-face inter-view with each participant in which the FSFI questions will be verbally asked and answered and compare between both groups in sexual activity and effect of chronic kidney disease on sexuality.

Duration of chronic kidney disease, duration of dialysis ,number of sessions of dialysis per week, medical treatment, haemoglobin,creatinine level will be fulfilled.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with chronic kidney disease stage 5 with estimated glomerular filtration rate (eGFR) <15 ml/min/1.7m2 using the equation of MDRD (modification of diet in renal disease) on dialysis or not.
* Age from 18 to 45 years old.
* Married.
* Sexually active during the last 6 months.

Exclusion Criteria:

* Pregnant women.
* Other medical diseases (diabetes mellitus, coronary artery disease, neurological disorders and other systematic diseases).
* Taking medications affect sexuality function e.g. antidepressant drugs.

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: The study will be conducted on 100 female patients divided in to two equal group:
  1. Group A: The patient group include 50 female patients with chronic renal failure (eGFR <15ml/min/1.7m2 )
  2. Group B: The control group including 50 healthy females age matched with the patient group.
  The Female Sexual Function Index (FSFI) will be used to assess sexual function. This index includes 19 questions related to 6 parameters: sexual desire, sexual arousal, lubrication, orgasm, sexual satisfaction and dyspareunia. A face-to-face inter-view with each participant in which the FSFI questions will be verbally asked and answered and compare between both groups in sexual activity and effect of chronic kidney disease on sexuality.
  Duration of chronic kidney disease, duration of dialysis, number of sessions of dialysis per week, medical treatment, haemoglobin, creatinine level will be fulfilled.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
evaluation of female sexual dysfunctions in patients with chronic kidney disease. | one year
  questionnaire to female patients with chronic kidney disease

CONTACTS AND LOCATIONS:
Locations (1):
- Esraa Ahmed Mohamed, Asyut, Egypt